CLINICAL TRIAL: NCT01735396
Title: A Pilot Study of Abiraterone Acetate in African American/Black Patients With Castration Resistant Prostate Cancer
Brief Title: Abiraterone Acetate Trial in African American Prostate Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: poor accrual
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Matthew Galsky, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-1727
Record Dates: First submitted 2012-11-24; First posted 2012-11-28 (Estimated); Results first posted 2017-05-12 (Actual); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: African American men; metastatic prostate cancer; castration resistant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abiraterone Acetate (Experimental): Abiraterone acetate 1000mg orally daily until the time of disease progression, in the absence of prohibitive toxicities.
  Interventions: Drug: Abiraterone Acetate

INTERVENTIONS:
Drug: Abiraterone Acetate — Abiraterone acetate 1000 mg orally daily (supplied as four 250 mg tablets) and prednisone 5 mg orally twice daily
  Other Names: Zytiga

SUMMARY:
This is a pilot study of abiraterone acetate in African American/Black patients with castration-resistant prostate cancer. The primary objective is to determine the correlation between germline polymorphisms and antitumor activity (as defined by a decline in PSA of ≥ 30%) in African American patients with castration-resistant prostate cancer treated with abiraterone acetate. Patients will receive abiraterone acetate until the time of disease progression, in the absence of prohibitive toxicities. Patients will be followed for disease progression and survival.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have signed an informed consent document indicating that the subjects understands the purpose of and procedures required for the study and are willing to participate in the study
* Be willing/able to adhere to the prohibitions and restrictions specified in this protocol
* Written Authorization for Use and Release of Health and Research Study Information
* African American or Black (by self identification)
* Male aged 18 years and above
* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Metastatic disease documented by standard imaging
* Progressive prostate cancer based on either rising PSA, new bone metastases, or progression of measurable disease according to PCWG2 12 guidelines.
* Patients in either of the following clinical states will be eligible for enrollment:

  i. No prior chemotherapy; ii. Patients previously treated with 1-2 prior chemotherapy regimens permitted, one of which must have been included docetaxel
* Surgically or medically castrated, with testosterone levels of < 50 ng/dl.
* Patients previously treated with an anti-androgen must demonstrate progression off of the anti-androgen.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 2
* Have a baseline serum potassium of ≥ 3.5 mEq/L
* Have aspartate aminotransferase (AST), alanine aminotransferase (ALT), and bilirubin levels < 1.5 x ULN
* Have a serum albumin of ≥ 3.0 g/dL
* Total bilirubin ≤ 1.5 x ULN
* Have a platelet count of ≥ 100,000/μL
* Have an absolute neutrophil count of > 1500 cell/mm3
* Have a calculated creatinine clearance ≥ 60 mL/min
* Have a hemoglobin of ≥ 9.0 g/dL
* Able to swallow the study drug as a whole tablet
* Willing to take abiraterone acetate on an empty stomach; no food should be consumed at least two hours before and for at least one hour after the dose of abiraterone acetate is taken
* Patients who have partners of childbearing potential must be willing to use a method of birth control with adequate barrier protection as determined to be acceptable by the principal investigator during the study and for 1 week after last dose of abiraterone acetate

Exclusion Criteria:

* Active infection or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated
* Known brain metastasis
* Uncontrolled hypertension (systolic BP ≥ 160 mmHg or diastolic BP ≥ 95 mmHg) Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III-IV heart disease or cardiac ejection fraction measurement of < 50% at baseline
* Administration of an investigational therapeutic within 30 days of screening
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements
* Have poorly controlled diabetes
* Have a history of gastrointestinal disorders (medical disorders or extensive surgery) that may interfere with the absorption of the study agents
* Have a pre-existing condition that warrants long-term corticosteroid use in excess of study dose
* Have known allergies, hypersensitivity, or intolerance to abiraterone acetate or prednisone or their excipients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Queens Cancer Center, Queens Hospital, New York, New York

REFERENCES:
- [Derived] Tsao CK, Sfakianos J, Liaw B, Gimpel-Tetra K, Kemeny M, Bulone L, Shahin M, Oh WK, Galsky MD. Phase II Trial of Abiraterone Acetate Plus Prednisone in Black Men With Metastatic Prostate Cancer. Oncologist. 2016 Dec;21(12):1414-e9. doi: 10.1634/theoncologist.2016-0026. Epub 2016 Oct 14. PMID 27742908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in Dec 2012, with enrollment from April 2014 to March 2016.
Period: Overall Study
Arm/Group | Abiraterone Acetate
Started | 11
Completed | 10
Not Completed | 1
Not completed — not evaluable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 66 [54 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Number of prior systemic therapies [Median (Full Range); unit: prior therapies] | 3 [1 to 4]
Performance Status: ECOG [Count of Participants; unit: Participants] — ECOG (Eastern Cooperative Oncology Group) Performance Status:
  0= Fully active; 1=restricted in physically strenuous activity but ambulatory, light work; 2= ambulatory and capable of self care, but no any work activities; 3= capable of only limited self care; 4 = completely disabled, 5= dead
  Participants
    ECOG 0 | 8
    ECOG 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With ≥ 30% Change in PSA
Description: The primary objective of this study is to determine a correlation between inherited genetic polymorphisms and antitumor activity (as defined by a decline in PSA of ≥ 30%) in AA patients with castration-resistant prostate cancer treated with Abiraterone. The primary endpoint is the percent change in PSA from baseline to 12 weeks. A decline of ≥ 30% will be correlated with germline SNPs.
Time Frame: baseline and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 10
Participants | 9

2. Secondary Outcome: Response Assessment
Description: Post-treatment changes in measurable disease by RECIST - Response Evaluation Criteria in Solid Tumors Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 10
Participants
  PR | 9
  SD | 1

3. Secondary Outcome: Time to Progression
Description: post-treatment changes in measurable disease by time to disease progression (as per PCWG2 guidelines)
Time Frame: up to 12 weeks
Population: data not collected
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 0

4. Secondary Outcome: Bone Scan
Description: post-treatment changes in bone scans (as per PCWG2 guidelines) ("no new lesions" versus "new lesions.")
Time Frame: up to 12 weeks
Population: data not collected
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 0

5. Secondary Outcome: Safety of Abiraterone
Description: To determine the safety of abiraterone Adverse events as defined by CTCAE v4. Number of participants with serious adverse events grade 4 or 5
Time Frame: up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 10
Participants | 0

6. Secondary Outcome: Testosterone
Description: Post-treatment changes in testosterone
Time Frame: up to 12 weeks
Population: data not collected
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Abiraterone Acetate
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=10)
Fatigue (General disorders) | 7
Hot flashes (General disorders) | 4
Nausea (General disorders) | 4
Vomiting (General disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Cough (General disorders) | 3
Alkaline phosphatase level increased (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Urinary incontinence (Renal and urinary disorders) | 3
Platelet count decreased (Blood and lymphatic system disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 5
Diarrhea (General disorders) | 2
Lymphocyte count decreased (Blood and lymphatic system disorders) | 4
Anorexia (General disorders) | 3
Muscle weakness in lower limb (Musculoskeletal and connective tissue disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Aspartate aminotransferase level increased (Metabolism and nutrition disorders) | 3
Alanine aminotransferase level increased (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes